CLINICAL TRIAL: NCT00001720
Title: Alendronate Versus Placebo for Idiopathic Juvenile Osteoporosis
Brief Title: Treatment of Childhood Osteoporosis With Alendronate (Fosamax)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980077; 98-CH-0077
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Osteoporosis
Keywords: Glucocorticoids; Bone Mineral Density; Bisphosphonates; Vertebral Fracture; Childhood Osteoporosis
MeSH Terms: conditions — Osteoporosis; Spinal Fractures | interventions — Alendronate

INTERVENTIONS:
Drug: Alendronate

SUMMARY:
Bones grow and stay strong through a continuous process of formation (building) and resorption (break down). When more bone is formed than resorbed, the density (level of calcium) in bone increases and the bones become stronger. However, if more bone is resorbed than formed the density of bone decreases and the bones become weak. This condition is called osteoporosis.

Osteoporosis is a rare but serious condition in children. Childhood osteoporosis can occur without a known cause (idiopathic juvenile osteoporosis). Children with osteoporosis suffer from pain, inability to stay active, and increased amounts of broken bones, including fractures of the spine. Even mild childhood osteoporosis may have long-term consequences since individuals who achieve a less than normal bone composition (peak bone mass) during the first 20-30 years of life may be at an increased risk for osteoporosis as adults.

Alendronate (Fosamax) is a drug that works by stopping bone resorption (break down). It has been used to treat post-menopausal osteoporosis, male osteoporosis and adults with osteoporosis due to long-term steroid therapy. The goal of this study is to determine the effectiveness of alendronate in children with idiopathic juvenile osteoporosis. Researchers believe that children treated with alendronate will improve bone strength and decrease the amount of fractures caused by osteoporosis.

DETAILED DESCRIPTION:
Osteoporosis is a rare but serious condition in children. One of the least well understood forms of childhood osteoporosis is idiopathic juvenile osteoporosis. Affected children suffer from pain, decreased activity tolerance, and increased fractures, including vertebral compression fractures. Even mild childhood osteoporosis may have long-term consequences since individuals who achieve a lower peak bone mass during the first 2-3 decades of life may be at increased risk for osteoporosis as adults.

Alendronate (Fosamax (Trademark), Merck & Co.), an aminobisphosphonate, is a potent inhibitor of bone resorption. It has been used to treat postmenopausal osteoporosis, idiopathic male osteoporosis, and glucocorticoid induced osteoporosis in adults. The goal of this protocol is to evaluate the effectiveness of Alendronate in children with glucocorticoid induced and idiopathic juvenile osteoporosis using a double-blind, randomized, placebo-controlled study design. We hypothesize that children treated with this drug will have an improvement in bone mineral density and decrease in osteoporotic fractures.

ELIGIBILITY:
INCLUSION CRITERIA:

Chronological age: 6.0 - 17.0 years. Study population will be restricted to children greater than 12 years of age until 8 patients have completed 6 months of the study or safety data is available from a comparable study.

AP Lumbar spine bone mineral density less than or equal to -2 standard deviations for age matched controls (z-score) using Hologic QDR machine.

Normative data published by Faulkner will be used to calculate Z-scores.

Patients with Idiopathic Juvenile Osteoporosis, osteoporosis (BMD less than -2 SD compared to age-matched controls) in a child with no identifiable etiology. Children with IJO and delayed puberty will have their z-score calculated on the basis of bone age.

EXCLUSION CRITERIA:

Inability to swallow pills or comply with administration instructions.

Upper gastrointestinal tract disease.

Creatinine clearance greater than or equal to 35 mL per min per 1.73 square meters.

Prior treatment with bisphosphonates.

Concurrent therapy with oral aspirin or salicylate containing compounds, excluding delayed-release salicylates which act in the distal gastrointestinal tract (for example, mesalamine, sulfasalazine, etc...).

Hypocalcemia.

Treatment with hGH or calcitonin in the preceding 6 months.

Inability to undergo dual energy x-ray absorptiometry.

Positive pregnancy test.

In females, sexual activity without an effective method of contraception.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1998-03; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bachrach LK. Bone mineralization in childhood and adolescence. Curr Opin Pediatr. 1993 Aug;5(4):467-73. doi: 10.1097/00008480-199308000-00017. PMID 8374675
- [Background] Brumsen C, Hamdy NA, Papapoulos SE. Long-term effects of bisphosphonates on the growing skeleton. Studies of young patients with severe osteoporosis. Medicine (Baltimore). 1997 Jul;76(4):266-83. doi: 10.1097/00005792-199707000-00005. PMID 9279333
- [Background] Falcini F, Trapani S, Ermini M, Brandi ML. Intravenous administration of alendronate counteracts the in vivo effects of glucocorticoids on bone remodeling. Calcif Tissue Int. 1996 Mar;58(3):166-9. doi: 10.1007/BF02526882. PMID 8852571